CLINICAL TRIAL: NCT05828407
Title: Fluid Challenge Impact in the Portal Vein Pulsatility Depending on the Fluid Responsivness Status
Acronym: FLUID-REVENGE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_1115; 2023-A00196-39 (Other: ID-RCB)
Record Dates: First submitted 2023-03-16; First posted 2023-04-25 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Insufficiency; Venous Congestion
Keywords: Point of care ultrasound; Portal vein pulsatility index; Venous congestion; Preload dependence
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Population:
  Critically ill patient with:
  * cardio circulatory insufficiency as defined by vasopressor requirement and at least one of the following criteria: arterial lactate >2mmol/L ; capillary refill time >3s ; mottling score >1 ; diuresis <0,5mL/h for more than 6hours
  * diameter of inferior vena cava >20mm
  Protocol:
  Administration of a fluid challenge (4mL/kg of Ringer Lactate) over 5 to 10 min.
  Point of care ultrasound evaluation of portal vein pulsatility index and Vexus criteria before and after the fluid challenge ; fluid challenge induced cardiac index variations estimated by pulse contour analysis

SUMMARY:
Portal vein pulsatility index is a marker of venous congestion evaluated by point of care ultrasound. It is associated with acute kidney injury, especially in critically ill patients. It may be considered as a dynamic marker. The investigators hypothesized that portal vein pulsatility index is higher after a fluid challenge only in patient without preload dependence in critically ill patients with cardiovascular insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* vasopressor requirement to maintain mean arterial pressure >65mmHg AND
* at least one of the following criteria:

  * arterial lactate >2mmol/L;
  * capillary refill time >3s;
  * mottling score >1;
  * diuresis <0,5mL/h for more than 6hours.

Exclusion Criteria:

* Diameter of vena cava <20mm
* Cirrhosis
* Pregnancy
* Severe acute pulmonary edema
* Phototype 4 or 5
* Patient opposition to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult intensive care patients with both grade 1 or higher venous congestion (VeXus C criteria) and acute circulatory failure.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Portal vein pulsatility index variation induced by the fluid challenge (%), defined by: Portal vein pulsatility index before the fluid challenge - portal vein pulsatility index after the fluid challenge. | One hour
  Portal vein pulsatility index is defined as the (maximal velocity - minimal velocity) / maximal velocity assessed with doppler in portal vein estimated with point of care ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Martin RUSTE, MD, Principal Investigator — Département d'anesthésie-réanimation
Locations (1):
- Hôpital cardiologique Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No